CLINICAL TRIAL: NCT00597298
Title: Randomized Controlled Trial on the Diaphragm Training With Threshold for Patient With Post-Cardiac Surgery Diaphragmatic Paralysis
Brief Title: Diaphragm Training Post-Cardiac Surgery
Acronym: DIATRACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedali Riuniti Trieste (Other)
Responsible Party: Marco Confalonieri/MD, SC Pneumologia - Ospedali RIuniti di Trieste
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: SCPN-01-08; PN 001-08
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Diaphragmatic Paralysis
Keywords: diaphragmatic paralysis; cardiac surgery; respiratory muscle training
MeSH Terms: conditions — Respiratory Paralysis | interventions — Speech Reception Threshold Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): inspiratory muscle training program using a pressure threshold device
  Interventions: Device: Threshold
- 2 (Sham Comparator)
  Interventions: Device: sham threshold

INTERVENTIONS:
Device: Threshold — Inspiratory muscle training program using a variable pressure device. An inspiratory muscle training device comprises a chamber having an opening for the passage of air to be inhaled and exhaled, and an inlet permitting air to be inhaled to enter the chamber and to pass to the opening. A one-way exhaust valve permits exhaled air entering through the opening to escape from the chamber, and another valve is provided to resist the entry of air to be inhaled into the chamber, the latter valve serving to vary the degree of resistance in dependence upon the volume of air that has passed through the inlet.
  Other Names: Threshold IMT, Respironics,Cedar Grove NJ, USA; HS730EU-010
  Arms: 1
Device: sham threshold — non-training physical activity
  Arms: 2

SUMMARY:
Diaphragm paralysis is a possible complication of cardiac surgery. The spontaneous recovery of the diaphragm mobility is slow and partial or absent in most cases. We hypothesize that a program of diaphragm muscle training by means of the Threshold variable resistance device could improve the rate of complete diaphragm mobility recovery in a shorter time period. Patient with post-cardiosurgical diaphragm paralysis will be random assigned to the specific training protocol or to a generic non-training physical activity.

DETAILED DESCRIPTION:
Inclusion criteria: All consecutive patients aged from 18 to 80 years old with RX-defined diaphragm paralysis post a major cardiosurgery intervention such as coronary bypass, valve substitution or both.

Exclusion criteria: Acute cardiac failure, COPD, chronic respiratory failure with indication to home oxygen therapy, neuromuscular diseases.

Outcome measures: MIP, MEP, diaphragm function recovery assessed by chest X-ray, lung function tests.

ELIGIBILITY:
Inclusion Criteria:

* post-cardiosurgical diaphragmatic paralysis recent cardiosurgical intervention for by-pass and/or valve replacement

Exclusion Criteria:

* heart failure
* COPD
* neuromuscular disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
chest x-ray mobility of the diaphragm | 6 and 12 months

SECONDARY OUTCOMES:
Maximal inspiratory pressure (MIP), cm H2O | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maja Demsar, MD, Study Director — AOUTS; Marco Confaloniei, MD, Study Chair — AOUTS
Locations (1):
- Fisiopatologia Respiratoria, Trieste, TS, Italy

REFERENCES:
- [Background] Versteegh MI, Braun J, Voigt PG, Bosman DB, Stolk J, Rabe KF, Dion RA. Diaphragm plication in adult patients with diaphragm paralysis leads to long-term improvement of pulmonary function and level of dyspnea. Eur J Cardiothorac Surg. 2007 Sep;32(3):449-56. doi: 10.1016/j.ejcts.2007.05.031. Epub 2007 Jul 19. PMID 17658265
- [Derived] Kodric M, Trevisan R, Torregiani C, Cifaldi R, Longo C, Cantarutti F, Confalonieri M. Inspiratory muscle training for diaphragm dysfunction after cardiac surgery. J Thorac Cardiovasc Surg. 2013 Mar;145(3):819-23. doi: 10.1016/j.jtcvs.2012.07.087. Epub 2012 Aug 29. PMID 22938776